CLINICAL TRIAL: NCT00517673
Title: A Two-Part Study to Evaluate Safety, Tolerability, and Pharmacokinetics of Single Escalating Oral Doses of GSK945237 and the Effect of Food on Single Oral Doses of GSK945237 in Healthy Adult Subjects
Brief Title: To Evaluate Safety, Tolerability, Pharmacokinetics, And Food Effect Of Single Doses Of GSK945237 In Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: BTI107248
Record Dates: First submitted 2007-08-15; First posted 2007-08-17 (Estimated); Last update posted 2012-03-19 (Estimated); Status verified 2011-10

CONDITIONS: Healthy Subjects; Infections, Bacterial
Keywords: Healthy Volunteer
MeSH Terms: conditions — Bacterial Infections | interventions — GSK945237; Sugars

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- GSK945237 (Experimental): Active Study Drug
  Interventions: Drug: GSK945237
- Sugar Pill (Placebo Comparator): Placebo
  Interventions: Drug: Sugar Pill

INTERVENTIONS:
Drug: GSK945237
  Arms: GSK945237
Drug: Sugar Pill — Placebo
  Arms: Sugar Pill

SUMMARY:
GSK945237 is the first molecule of a new chemical class that is being developed for treatment of respiratory tract and other infections such as skin and soft tissue. This study drug has been tested in animals but has never been given to humans. This is a two part study. The purpose of the first part is to study the side effects of this drug in humans, and to study how much of the drug gets absorbed in the blood stream The second part of this study will compare absorption of the study drug in the blood stream when given with food and when given under fasting conditions

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female adults between 18 and 60 years of age.
* Body weight proportional to height.
* Female subjects must be of non-childbearing potential.
* QTc less than 450 msec at screening

Exclusion Criteria:

* Any clinically relevant abnormality identified on the screening history and physical, or on laboratory evaluations or the 12-lead surface electrocardiogram at screening or pre-dose.
* A positive pre-study alcohol/urine drug screen.
* Use of nicotine-containing products.
* A positive pre-study HIV antibody, Hepatitis B surface antigen (HBsAg) or Hepatitis C antibody result.
* Recent participation in another study, use of certain medications, consumption certain fruits, juices, or red wine

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 68 (Actual)
Dates: Start 2007-07; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability | Day 1 to follow-up visit

SECONDARY OUTCOMES:
Pharmacokinetics | Day 1 to Day 5

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Adelaide, South Australia, Australia